CLINICAL TRIAL: NCT05060185
Title: A Prospective, Multicenter,Single Arm Clinical Investigation Evaluating Safety and Effectiveness of the Flow Diverter for Treating Patients With Intracranial Aneurysms
Brief Title: The Flow Diverter for Treating Patients With Intracranial Aneurysms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu CED Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CER-A-FD-01
Record Dates: First submitted 2021-09-14; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-08

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): the patients will be treated by the trial device
  Interventions: Device: the Flow Diverter

INTERVENTIONS:
Device: the Flow Diverter — Those who meet the inclusion criteria but do not meet the exclusion criteria will be enrolled through the electronic central registration system. The investigator log in to the central registration system, fill in the subject information and submit it who enroll in the study. The investigator complete the surgery and conduct relevant evaluation according to the protocol.

SUMMARY:
To evaluate the efficacy and safety of the blood flow guide device manufactured by Jiangsu Changyida Medical Technology Co., Ltd. for endovascular embolization of intracranial aneurysms

ELIGIBILITY:
Inclusion Criteria:

●≥18 years old and ≤75 years old, male or unpregnant female

* Untreated and unruptured intracranial wide-necked aneurysm confirmed by preoperative imaging diagnosis (wide-necked aneurysm was defined as the tumor neck ≥4mm or the tumor body/tumor neck ratio <2)
* The target aneurysm is planned to be treated with blood flow guidance device only, without the need to complete the treatment by stages
* The width of tumor neck should be less than 30mm
* Imaging measurements of the tumor parent artery showed that the diameter was 1.5mm ~ 6.5mm
* The subject or legal guardian can understand the purpose of the study, demonstrate sufficient compliance with the study protocol, and sign the informed consent

Exclusion Criteria:

* The target aneurysm has previously received craniotomy clipping or other endovascular interventional treatment
* Target aneurysms were haemacular aneurysms, pseudoaneurysms, arteriovenous malformations and moyamoya disease related aneurysms
* DSA suggested vascular path tortuosity or severe arteriosclerosis, and it was difficult for the instrument to reach the target vessel
* Contraindications to dual antiplatelet therapy and anticoagulation therapy
* Patients with known clear allergy to nickel-titanium alloys and platinum-tungsten alloys
* People with known severe allergy to contrast media (excluding rash)
* patients with known dementia or mental illness
* Preoperative complicated with serious heart, liver, kidney, respiratory system diseases and bleeding disorders
* Life expectancy is less than one year
* Is participating in, or may participate in, any other drug or medical device clinical trial after inclusion in this clinical trial
* Other conditions determined by the investigator to be unsuitable for participation in this clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-10-17 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The rate of complete aneurysm occlusion (Raymond score: Ⅰ) confirmed by 12 postoperative menstrual imaging | Twelve months after surgery
  The cerebral vascular imaging examination 12 months after the operation was performed to analyze whether the aneurysm was completely occluded. Aneurysm occlusion images were reviewed by clinicians and the core laboratory respectively. When the evaluation results were different from those determined by clinicians, the results of the core laboratory should prevail

SECONDARY OUTCOMES:
Immediate postoperative success rate | Immediately after
  The intraoperative blood flow guidance device was successfully released, and the implant was accurately located by angiography after placement, and the proportion of subjects who could effectively cover aneurysma neck was calculated.
The parent artery was unblocked 12 months after surgery (stenosis rate ≤50%) and no further intervention was performed | Twelve months after surgery
  The clinician and the core laboratory will evaluate the results respectively. If the evaluation results are different from those determined by the clinician, the core laboratory results shall prevail
The rate of self-care (mRS 0-2 points) at 12 months after operation | Twelve months after surgery
  MRS is a disability assessment to assess the independent living standard of postoperative patients and analyze the outcome of aneurysm surgery.